CLINICAL TRIAL: NCT04164368
Title: Lenalidomide Combined With R-CHOP in Newly Diagnosed Double-expressor Diffuse Large B-Cell Lymphoma Patients
Brief Title: Lenalidomide Combined With R-CHOP(R2-CHOP) in Newly Diagnosed Double-expressor Diffuse Large B-Cell Lymphoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junning Cao, MD, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DE-LYM2019
Record Dates: First submitted 2019-10-23; First posted 2019-11-15 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Double Expressor Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R2-CHOP (Experimental): Lenalidomide combined with rituximab, cyclophosphamide, vincristine, doxorubicin, prednisone
  Interventions: Drug: Lenalidomide combined with R-CHOP

INTERVENTIONS:
Drug: Lenalidomide combined with R-CHOP — rituximab 375 mg/m2,ivgtt D1 cyclophosphamide 750 mg/m2 iv D2 vincristine 1.4 mg/m2 [capped at 2.0 mg], iv D2 doxorubicin 50 mg/m2 iv D2 prednisone 100 mg/m2 per day PO D2-6 Lenalidomide 25mg PO QD D2-11
  Other Names: R2-CHOP

SUMMARY:
In this phase II study, the investigators are aiming to explore lenalidomide combined with R-CHOP (R2-CHOP) in newly diagnosed double-expressor Diffuse Large B-Cell Lymphoma patients (DLBCL)

DETAILED DESCRIPTION:
Double expressor lymphoma is a subtype of diffuse large B-cell lymphoma defined as having increased expression of MYC and BCL-2 by immunohistochemistry. Patients with double-expressor lymphomas have a poor prognosis when treated with standard chemoimmunotherapy and have increased risk of progression and recurrence. The investigators conducted this study to evaluate the efficacy of lenalidomide combined with R-CHOP (R2-CHOP) in newly diagnosed double-expressor, untreated Diffuse Large B-Cell Lymphoma patients (DLBCL). Lenalidomide is the second-generation immunomodulatory drug, and its anti-tumor mechanism may involve immunomodulatory, antiinflammatory, and antiangiogenic effects and suppression of tumor necrosis factor-alpha (TNF-α) from peripheral blood mononuclear cells. In this phase II study, the investigators are aiming to explore lenalidomide combined with R-CHOP (R2-CHOP) in newly diagnosed double-expressor Diffuse Large B-Cell Lymphoma patients (DLBCL), in order to find a potential promising way to treat this kind of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-75 years old
2. Eastern Cooperative Oncology Group performance status 0 to 2;
3. Newly diagnosed, untreated, histological confirmed diffuse large B cell lymphoma, and Myc≥40% as well as Bcl-2≥50% through immunohistochemistry；
4. Measurable disease was defined as at least one lesion ≥1.5 cm in length-diameter and ≥1.0cm in short-diameter by CT or MRI.
5. White blood cell ≥ 3.5×109/L, absolute neutrophil count ≥ 1.5×109/L，platelet ≥ 80×109/L，hemoglobin ≥ 90 g/L. If abnormal factors of peripheral blood caused by bone marrow or spleen involvement of lymphoma, whether to enroll depends on the judgment of researchers
6. Total bilirubin < 1.5×upper limit of normal(ULN), ALT and AST < 1.5× ULN
7. serum creatine <1.5×ULN, and creatinine clearance rate (CCR) ≥ 40 ml/min
8. Ultrasonic cardiogram or nuclide cardiac function showed left ventricle ejection fraction ≥ 50%
9. Women of childbearing potential and men who are sexually active are consent to practicing a highly effective method of birth control. Women of childbearing potential must have a negative serum β-hCG within 2 weeks of enrollment
10. Patients have written informed consent to participate in the study.

Exclusion Criteria:

1. Prior sever allergy to humanized or mouse derived monoclonal antibody. Unable to receive either lenalidomide or R-CHOP background chemotherapy.
2. History of myocardial diseases, such as unstable angina pectoris, acute myocardial infarction within 6 months of enrollment, congenital heart failure NYHA III/IV
3. Particular kind of DLBCL，such as primary mediastinal/thymic B-cell lymphoma, EBV positive DLBCL, primary cutaneous large B lymphoma, leg type.
4. Presence of CNS involvement
5. Having surgeries ≥ grade 2 within 3 weeks of enrollment.
6. History or now in the treatment process of other malignancies except cured basal cell carcinoma of skin (melanoma not included), and carcinoma in-situ of uterine cervix.
7. More than grade 3 neurotoxicity within 2 two weeks of enrollment
8. Receiving any treatment for lymphoma except short use of corticosteroid (no more than 10 days)
9. History of deep vein thrombosis or pulmonary embolism within 12 months of enrollment
10. Unable or reject to receive antithrombotic treatment
11. Presence of active HBV infection (HBsAg positive and HBV-DNA≥ 104), HCV infection, acquired and congenital immunodeficiency diseases include but not limited to HIV
12. Pregnant or lactating women
13. Previously received organ transplant
14. Serious uncontrolled infection
15. Having contraindications to the use of large doses of hormone, such as uncontrolled hyperglycemia, gastric ulcer, mental disorder.
16. Severe neurol of mental illness, including dementia and epilepsy.
17. Drug abuse, medical, psychological or social conditions which may interfering with subjects' participation in the study or evaluation of the results
18. Patients considered unsuitable to participate in the study by the researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
2-year progression free survival | From date of patients sign informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed progression of the disease or the occurrence of death for any reason

SECONDARY OUTCOMES:
objective response rate | at the end of Cycle 6 (each cycle is 21 days)
  the ratio of numbers of patients with complete response and partial response to all the participants receiving treatment
overall survival | From date of patients sign informed consent until the date of death or the date of last follow-up time, whichever came first, assessed up to 2 years
  time between the date of patients sign informed consent and the date of death or the date of last follow-up time
Hematology and non hematology toxicity | Throughout the treatment period，up to 6 months
  number of participants with treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
serum cfDNA biomarkers and tissue biomarkers | up to 2 years
  detection of serum and tissue biomarkers in the treatment of double-expressor lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Junning Cao, Principal Investigator — Fudan University
Locations (1):
- 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No